CLINICAL TRIAL: NCT01265914
Title: A Randomised, Double-Blind, Placebo-Controlled, Ascending Dose Study to Assess the Safety, Tolerability and Immunogenicity of Repeated Intramuscular Administration of an Influenza A Vaccine (FP-01.1)
Brief Title: A Study to Evaluate the Safety, Tolerability and Immunogenicity of a Universal Influenza A Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immune Targeting Systems Ltd (Industry)
Collaborators: Hammersmith Medicines Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FP-01.1_CS_01
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Biological: placebo
- FP-01.1 (Experimental)
  Interventions: Biological: FP-01.1

INTERVENTIONS:
Biological: FP-01.1 — Ascending doses of FP-01.1 will be administered
  Arms: FP-01.1
Biological: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and immunogenicity of ascending doses of a novel, universal flu vaccine, in healthy volunteers.

DETAILED DESCRIPTION:
FP-01.1 is composed of a mixture of synthetic peptides, modified with a fluorocarbon vector, which is anticipated to enhance the immune properties of the drug, and allows differentiation from recent investigational interventions by avoiding the use of adjuvant. The peptide sequences, derived from internal influenza-A proteins, were selected based on the presence of CD4+ and CD8+ T cell epitopes and a high degree of conservation across all influenza strains, using a proprietary bioinformatics approach, and, it is proposed, will enable FP-01.1 to universally treat influenza-A -infected populations.

This study is the initial exploration of the safety, tolerability and immunogenicity response of FP-01.1 in healthy volunteers. Ascending doses of FP-01.1 will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 55 years inclusive at the time of consent
2. Male and female subjects who are willing to comply with the applicable contraceptive requirements of the protocol
3. Satisfactory medical assessment with no clinically significant or relevant abnormalities in medical history, physical examination, vital signs, ECG and laboratory evaluation (haematology, biochemistry or urinalysis) as assessed by the Investigator.
4. Ability to provide written, personally signed and dated informed consent to participate in the study.
5. The subject has a body mass index within the range 19.0-32.0 kg/m2 and falls within the weight range of 50.0-100.0 kg.
6. Subject is willing to refrain from consuming alcohol for 24h prior to all visits.

Exclusion Criteria:

1. As a result of the medical screening process, the Principal Investigator or Co-Investigator considers the subject unfit for the study.
2. Current or recurrent disease (e.g. cardiovascular, respiratory, endocrine, renal, liver, gastrointestinal, autoimmune, immune suppression, malignancy or other conditions) that could affect the action, absorption or disposition of the investigational medicinal product (IMP) or could affect clinical or laboratory assessments.
3. Significant illness as judged by the Principal Investigator or Co-Investigator within 2 weeks of the first dose of IMP.
4. Subjects with a history of allergies or allergic conditions including asthmatics, hay fever and eczema sufferers requiring medication which in the opinion of the Principal Investigator or Co-Investigator will affect their participation in the study.
5. Concurrent use of any medication (including prescription, over the counter, herbal or homeopathic preparations and any vaccinations (including travel vaccinations).
6. Known or suspected intolerance or hypersensitivity to the IMP/placebo, or closely related compounds or any of the stated ingredients.
7. History of alcohol or other substance abuse within the last year. A positive screen for alcohol or drugs of abuse.
8. Male subjects who consume more than 21 units of alcohol per week and female subjects who consume more than 14 units of alcohol per week.
9. A positive HIV antibody screen, Hepatitis B surface antigen, Hepatitis B core antibody, or Hepatitis C antibody screen
10. Subjects who have significant scarring, tattoos, abrasions, cuts or infections at the dose site that in the opinion of the Investigator could interfere with evaluation of injection site local reactions.
11. Donation of blood or blood products (e.g. plasma, platelets) within 90 days prior to or intention to donate blood during the entire study.
12. Use of another investigational medicinal product within 90 days prior to receiving the first dose of IMP or intention to enrol in another clinical study throughout the entire study including the follow up period.
13. Subject with suspected recent (≤12 months) pre-exposure to the influenza A virus
14. Subjects who have received a flu vaccine in the last 12 months or who anticipate receiving it within the duration of the study including follow up.
15. Any clinically significant abnormalities, in the opinion of the Principal Investigator or Co-Investigator, on electrocardiograms

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

SECONDARY OUTCOMES:
Immunogenicity of FP-01.1.
  Immunogenicity of ascending doses will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Steve Warrington, MD, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research Ltd, London, United Kingdom

REFERENCES:
- [Derived] Francis JN, Bunce CJ, Horlock C, Watson JM, Warrington SJ, Georges B, Brown CB. A novel peptide-based pan-influenza A vaccine: a double blind, randomised clinical trial of immunogenicity and safety. Vaccine. 2015 Jan 3;33(2):396-402. doi: 10.1016/j.vaccine.2014.06.006. Epub 2014 Jun 10. PMID 24928790